CLINICAL TRIAL: NCT03539523
Title: Investigation of the Validity and Reliability of the L Test in Children With Cerebral Palsy
Brief Title: L Test in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Sebahat Yaprak Cetin, Principal investigator, Pamukkale University
Other Study IDs: 60116787-020/78784
Record Dates: First submitted 2018-05-16; First posted 2018-05-29 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Cerebral Palsy
Keywords: L test; cerebral palsy; children; validity; reliability
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to investigation of the validity and reliability of the L test in children with cerebral palsy. Eighty children with CP with mean age of 11.60±3.85 (56 boys, 24 girls) were included in the study. ICC ((Intraclass Correlation Coefficient) was used to assess interclass, intraclass and test- retest validity of the L test. Two independent examiners made L test, for the inter-rater reliability, twice within 1 day for the test-retest reliability. The minimal clinical important difference at 95% confidence interval intra-class correlation coefficient and standard error of measurements were calculated. The correlations of L test with Timed up and Go Test (TUG) and Timed up and Down Stairs Test (TUDS) were assessed for concurrent validity.

DETAILED DESCRIPTION:
Inclusion criteria were: cerebral palsy diagnosis, absence of other diseases that may impact gait performance, ambulatory for at least 20 meters, maximum level 2 according to Gross Motor Function Classification System. Exclusion criteria were: difficulty in following the instructions, severe lower extremity pain that affects mobility, orthopedic surgery within the last 12 months, Bothulium toxin A injection for lower extremity within the last 3 months and walking with a physical assistance from another person. Informed consents were obtained from the parents of the participants for the trial. Assessments were conducted in a special training and rehabilitation center where children with cerebral palsy received regular treatments.

ELIGIBILITY:
Inclusion Criteria:

* cerebral palsy diagnosis, absence of other diseases that may impact gait performance, ambulatory for at least 20 meters, maximum level 2 according to Gross Motor Function Classification System

Exclusion Criteria:

* difficulty in following the instructions, severe lower extremity pain that affects mobility, orthopedic surgery within the last 12 months, Bothulium toxin A injection for lower extremity within the last 3 months and walking with a physical assistance from another person.

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2018-01-02 (Actual); Study Completion 2018-04-02 (Actual)

PRIMARY OUTCOMES:
L test | 1 hour
  The child sat down on a armchair with their back on the backrest, then got up from the chair with the start command, walked the L-shaped 10 meters (3m+7m), turned back, walked the same distance and sat down the chair again. Time lapsed was recorded in seconds

SECONDARY OUTCOMES:
Timed Up and Go test | 10 minutes
  The child got up from the chair with the start command, walked for 3 meters, turned around, walked back and sat down. The time between the start command and the moment of complete seated position was recorded in seconds

OTHER OUTCOMES:
Timed Up and Down Stairs test | 10 minutes
  A 10-step ladder was used for this test. The child was asked to climb up to the step at the top with the start command, turn back and climb down.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Kınıklı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
Shared during work writing

REFERENCES:
- [Result] Nguyen VC, Miller WC, Asano M, Wong RY. Measurement properties of the L test for gait in hospitalized elderly. Am J Phys Med Rehabil. 2007 Jun;86(6):463-8. doi: 10.1097/PHM.0b013e31805b8193. PMID 17515685
- [Result] Deathe AB, Miller WC. The L test of functional mobility: measurement properties of a modified version of the timed "up & go" test designed for people with lower-limb amputations. Phys Ther. 2005 Jul;85(7):626-35. PMID 15982169